CLINICAL TRIAL: NCT04593992
Title: High-tone External Muscle Stimulation for Treatment of Diabetic Polyneuropathy
Brief Title: HTEMS Treatment of Diabetic Polyneuropathy
Acronym: HTEMS-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Collaborators: gbo Medizintechnik AG (Unknown)
Responsible Party: Principal Investigator, Stephan Martin, Principal investigator, West German Center of Diabetes and Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP study
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diabetic Polyneuropathy
Keywords: diabetes; neuropathy; pain; HTEMS
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HTEMS (Experimental): High-tone external muscle stimulation 5 times within a week for 12 weeks
  Interventions: Device: HTEMS
- Placebo (Placebo Comparator): Placebo stimulation 5 times within a week for 12 weeks
  Interventions: Device: Placebo

INTERVENTIONS:
Device: HTEMS — high-tone external muscle stimulation
  Other Names: HITOP 191 (gbo Medizintechnik AG, Rimbach, Germany)
  Arms: HTEMS
Device: Placebo — Placebo stimulation
  Other Names: Placebo treatment
  Arms: Placebo

SUMMARY:
So far, there are no sufficient pharmacologic therapies for the treatment of diabetic neuropathy. Therefore, we evaluated application of high-tone external muscle stimulation (HTEMS) compared to placebo treatment in patients with diabetic neuropathy.

DETAILED DESCRIPTION:
Patients (n=80) with symptomatic diabetic neuropathy will be included into this randomized controlled trial. Each intervention will be administered for a period of at least 30 min on at leat 5 days in a week. Health impairments will be assessed using the neuropathy symptom score (NSS) before, during and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic diabetic neuropathy
* stable oral analgesic regimen

Exclusion Criteria:

* history of drug or alcohol abuse
* cardiac pacemaker or defibrillator
* pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Neuropathy symptom score | 12 weeks
  Neuropathic symptoms measured by the neuropathic symptom score (NSS). Range 1-10 with higher scores indicationg a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- West-German Centre of Diabetes and Health, Düsseldorf Catholic Hospital Group, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No